CLINICAL TRIAL: NCT03281980
Title: Effects of Adding Psychosocial Stimulation for Children of Lactating Mothers Enroled to Receive Unconditional Cash Transfer (UCT) and Health Education Awareness Programme on Children's Cognition and Behaviour in Rural Bangladesh
Brief Title: Effects of Psychosocial Stimulation and Cash on Children's Development and Behaviour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR-17009
Record Dates: First submitted 2017-08-17; First posted 2017-09-13 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-02

CONDITIONS: Child Development; Child Behavior
Keywords: Bangladesh; Child development; Poor mothers; Psycho social stimulation; Unconditional cash transfer
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The testers of the participants will not have the information about type of intervention of the children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (UCT+HE+PS) (Experimental): The participants of this arm will receive UCT and HE along with psychosocial stimulation (PS)
  Interventions: Other: Psychosocial stimulation (PS)
- Government Intervention (UCT+HE) (Sham Comparator): The participants of this arm will receive only UCT and HE
  Interventions: Other: Government Intervention (UCT+HE)
- Comparison (No Intervention)

INTERVENTIONS:
Other: Psychosocial stimulation (PS) — i) Unconditional Cash Transfer(UCT)/ Maternity Allowance: MoWCA, GoB provides maternity allowance of taka 500 ($6.25) for each mother up to two years in each month.
  ii) Health Education Awareness Program: All mothers receive health education training by designated LNGOs/CBOs
  iii) Psychosocial stimulation: The participants will receive fortnightly sessions at home.
  Arms: Intervention (UCT+HE+PS)
Other: Government Intervention (UCT+HE) — fgbfgjhgykghilk
  Arms: Government Intervention (UCT+HE)

SUMMARY:
Burden: In developing countries, an estimated 219 million children do not reach their maximum potentiality because of poverty and associated risk factors. More than half of the Bangladeshi children <5 years are at risk for developmental delay due to poverty and sub-optimal home stimulation. Sometimes poor people become poorer due to catastrophic expenditure on health care and fall into the vicious cycle of poverty

Knowledge gap: Although, there is evidence that conditional cash transfer helps develop poor people' health and nutritional status, little is known about the effect of unconditional cash transfer and health education (HE) programmes along with psychosocial stimulation on children' cognition and behaviour.

Relevance: The study will bring an opportunity to evaluate the effect of transferring unconditional cash and health education programme along with psychosocial stimulation to poor families under safetynet programme of Bangladesh Govt. in rural areas. The study will also document direct and indirect cost to measure cost effectiveness that will help in decision making to implement the project if it shows benefits to children's development.

Primary Hypothesis (if any):

* Unconditional cash transfer (UCT) and health education (HE) programme will improve child's cognitive, motor and language development and behaviour compared to no intervention group.
* Adding psychosocial stimulation to an unconditional cash transfer (UCT) and health education (HE) programme will will have an additive effect on Childs's cognitive, motor and language development and behaviour compared to the control groups

Secondary Hypothesis:

Additionally the intervention will

* be cost effective,
* reduce mothers' depressive symptoms and improve their self esteem
* improve children's growth and household food security status
* reduce domestic violence
* Health seeking behaviour and health care expenditure

Long-term goal: our ultimate goal is to find a suitable infrastructure to take to scale early child development activities for the whole country.

Methods: It is a Cluster Randomized Controlled Trial with three-arms (i) UCT+HE+Psychosocial stimulation (ii) UCT+HE and iii) Comparison group.

DETAILED DESCRIPTION:
Primary objectives:

To evaluate the effect of UCT and HE programme on children's cognitive, motor and language development and behaviour To evaluate the effect of adding psycho social stimulation to an UCT and HE program on cognitive development and behavior of young children

Secondary objectives are:

To measure effect of the program on:

cost effectiveness of the intervention mothers'mental health (depression symptoms) and their self esteem household food security status and children's growth and domestic violence health care expenditure and health seeking behaviour of the families

Introduction:

In developing countries, an estimated 250 million children younger than 5 years in low and middle income countries do not reach their maximum potentiality because of poverty and associated risk factors. More than half of the Bangladeshi children less than 5 years are at risk for developmental delay due to poverty and sub-optimal home stimulation. Sometimes poor people become poorer due to catastrophic expenditure on health care and fall into the vicious cycle of poverty. Conditional and unconditional cash transfer to the poor mothers has proved a way of reducing poverty and improving health outcomes for mothers and children worldwide. Ministry of Women and Children Affairs (MoWCA),Government of Bangladesh (GoB) introduced maternity allowance in the fiscal year 2007-2008. This is an unconditional cash transfer under safety net program for the poor mothers. The mothers also receive health education awareness program. The overall objective of the cash and health education training program is to ensure safety net in terms of morbidity, mortality and welfare during pregnancy and lactation period for both mother and child. Adding psycho social stimulation to the program will benefit children's cognition, behavior and nutritional status. On the other hand the interventions together will address family's food security and mothers' physical and mental health and self esteem because receiving extra cash as well as education on health and psycho social stimulation will enhance mothers' capacity in many aspects.

Psycho social stimulation alone and along with other health and nutrition programs was found to be effective for children's cognition and behavior [9-13]. Conditional Cash Transfer (CCT) alone was also found significantly effective for child development in Mexico. On the other hand, studies reported that UCT improved other health outcomes and nutrition, but little is known about the effect of unconditional cash transfer (UCT) along with health education program and psycho social stimulation on children's cognition and behavior. MoWCA is transferring cash to poor pregnant mothers along with health education training program under social safety net program. The present study group plan to conduct a randomized controlled trial to document effect of adding psycho social stimulation to the present program on children's cognition and behavior. 200 mother-child dyads in each arm will be enrolled when their child is 6-16 months old. The participants of the intervention group will receive psycho social stimulation fortnightly at home for 12 months.

However, UCT and HE program is a social safety net program under the ministry of Women and Children Affairs of Bangladesh Government. The outcomes of this program are primarily maternal and child health and does not directly focus on children's cognition and behavior. However, social safety net programs may indirectly affect other outcomes like maternal depressive symptom, violence against women, children's well being, cognition and behavior and nutrition status for both mother and child. The researchers intend to add psycho social stimulation in order to trigger the outcomes in terms of children's development. But the program needs to be cost effective to be scale able in low resources settings. If the intervention is cost effective, the package may be found attractive by respective policy makers to improve development of poor children in those settings.

The maternity allowance of taka 500 ($6.25) per month is distributed through commercial banking system. Health education awareness program is conducted monthly by some Local Non Government Organizations (LNGOs) and Community Based Organizations (CBOs) on a wide range of health and social welfare issues. The NGO,/CBOs have their own curriculum approved by MoWCA for the awareness program. The Local government and community leaders can play an important role in encouraging the eligible women to participate in the program. Home based psycho social stimulation will be provided by community female Play leaders having at least 12 years of education. So the project will build capacity of the community including the Play Leaders from the community.

Study design:

This is a cluster randomized controlled trial with 3 arms: i) Psychosocial stimulation+ Health education program + Unconditional cash transfer ii) Health education program + Unconditional cash transfer and iii) Comparison arm. The comparison group will consist of those who are eligible to receive UCT but do not receive it due to resource constraints of the UCT programme.

Recruitment:

11 Unions have been selected randomly out of 14 Union at Ullapara, a sub district under Sirajgonj district in Bangladesh.The old Ward of a Union would be considered as cluster.

Since the Government is providing UCT to 79 mothers in each Union, the research team assume to get approximately 26 participants in each Ward. 18 participants will be enrolled randomly from each cluster. Restricted randomization process will be followed. There are three old Wards in each Union. the each old ward (cluster) will be allocated for each arm randomly.

For comparison arm, mother-child dyads will be enrolled from any part of the old Ward until the required sample size are fulfilled.The eligibility criteria of participants for the comparison arm would be the same as that for the UCT recipients.

Intervention and Project Execution Plan:

The study aims to integrate three distinct interventions: i) Maternity allowance ii) Health education awareness program and iii) Psychosocial stimulation.

i) Maternity Allowance: MoWCA, GoB provides maternity allowance of taka 500 ($6.25) for each poor pregnant mother up to two years through banking channel under safety net program of the GoB.

ii) Health Education Awareness Program: All mothers receiving maternity allowance receive various health education training by designated LNGOs/CBOs through MoWCA, GoB funding.

iii) Psychosocial stimulation: The participants will receive fortnightly sessions of psychosocial stimulation at home by community female play leaders for one year. The curriculum of stimulation is based on improving the mother-child interaction, and providing developmentally appropriate activities for the child. The curriculum has already been used in several projects in Bangladesh run by Child Development Unit of icddr,b and has shown significant benefits to children's development[10-12, 22] and growth[11, 22].

Training:

When the inter observer reliability coefficient will be more than 0.8 through data collection training, will be considered that the trainee to be eligible to take part in the test procedure. Quality of data collection will be checked at the field by supervisors/master trainers on 10% of the assessments.

Data collection:

All data will be collected from all groups- Group I: UCT+HE Group II: (UCT+HE)+ Psychosocial stimulation and group III: Comparison. Data will be collected at baseline, end line and some others monthly to compare the outcome between the groups.

Data Storage Data will be stored in databases saved on icddr,b servers.The databases will be password protected and only members of the study team and investigators will have access to the password.

Sample size The study requires 200 mother-child dyads in each arm with 11 clusters of 18 participants in each cluster. So in total we will have 600 participants, 33 cluster, 18 participants in each cluster considering 90% power, 5% level of significance, an intraclass correlation (ICC) of 0.05 and an effect size of previous study.

Data analysis:

Data will be checked for normality. Appropriate measures will be taken if there are any abnormal distributions. Differences between groups in socioeconomic and other background characteristics will be analyzed using t-test for continuous variables for two groups and a ANOVAforthree groups. Effect of the interventions will also be measured using intention-to-treat analysis controlling for the clustering effect.

.

Cost-effectiveness Analysis:

The objective of the study is to estimate the resources used and costs associated with interventions. The research team will measure direct and indirect cost of for all the groups. Average costs per participants will be calculated by multiplying the cost of resource items by their respective unit costs. The outcomes of the study will be measured. Then the incremental cost-effectiveness ratio (ICER) will be used in cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a child aged 6-16 months
* Eligible to receive UCT.

  * UCT+HE+PS arm: Receiving unconditional cash from government
  * UCT+HE arm: Receiving unconditional cash from government
  * Comparison arm: eligible to receive UCT but not under UCT programme.
* Not expected to leave the study site for more than 2 months
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* Legal guardian unwilling or unable to provide written informed consent.
* Known congenital anomaly
* Developmental disorder or severe developmental delay
* Not possible to test the child due to physical or behavioral problems
* Children of multiple birth e.g. twin, triplets

Ages: 6 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Child development composite score | Change children's cognition, language and motor as composite score after one year intervention
  Children's cognition, language and motor as composite score
Children's behavior and composite score | Change children's behaviour after one year intervention
  Children's behavior will be measured by Wolk's behavior rating scale during bayley

SECONDARY OUTCOMES:
Children's weight | Change children's weight after one year intervention
  Children's weight will be measured by Gram
Children's height | Change children's height after one year intervention
  Children's height will be measured by centimeter
Children's Mid Upper Arm circumference (MUAC) | Change children's MUAC after one year intervention
  Children's MUAC will be measured by millimeter
Mothers' weight | Change mother's weight after one year intervention
  Mothers' weight will be measured by Gram
Mothers' height | Change mother's height after one year intervention
  Mothers' height will be measured by Centimeter
Mothers' depressive symptom | Change mother's depression status after one year intervention
  Mothers' depressive symptom will be measured by Self-Regulation Questionnaire (SRQ)
Mothers' level of self-esteem | Change mother's level of self esteem after one year intervention
  Mothers' level of self-esteem will be measured by Rosenberg Self-esteem questionnaire
Family's monthly food security status | Change family's food security status after one year intervention
  Family's monthly food security status will be measured by Household Food Insecurity Access Scale (HFIAS) questionnaire
Family's monthly health seeking behavior | Change family's health seeking behaviour status after one year intervention
  Family's monthly health seeking behavior status will be measured by questionnaire
Family's monthly income | Change family's income status after one year intervention
  Family's monthly income status will be measured by questionnaire
Family's monthly expenditure | Change family's expenditure status after one year intervention
  Family's monthly expenditure status will be measured by questionnaire
Domestic violence (mothers) | Change family's domestic violence status after one year intervention
  Domestic violence (mothers) monthly status will be measured by questionnaire
Family care indicators (FCI), | Change of FCI after one year intervention
  Family care indicators (FCI) will be measured by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Upazilla, Sirajganj, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Background] Hamadani JD, Tofail F, Hilaly A, Huda SN, Engle P, Grantham-McGregor SM. Use of family care indicators and their relationship with child development in Bangladesh. J Health Popul Nutr. 2010 Feb;28(1):23-33. doi: 10.3329/jhpn.v28i1.4520. PMID 20214083
- [Background] Hamadani JD, Tofail F, Huda SN, Alam DS, Ridout DA, Attanasio O, Grantham-McGregor SM. Cognitive deficit and poverty in the first 5 years of childhood in Bangladesh. Pediatrics. 2014 Oct;134(4):e1001-8. doi: 10.1542/peds.2014-0694. PMID 25266433
- [Background] van Doorslaer E, O'Donnell O, Rannan-Eliya RP, Somanathan A, Adhikari SR, Garg CC, Harbianto D, Herrin AN, Huq MN, Ibragimova S, Karan A, Ng CW, Pande BR, Racelis R, Tao S, Tin K, Tisayaticom K, Trisnantoro L, Vasavid C, Zhao Y. Effect of payments for health care on poverty estimates in 11 countries in Asia: an analysis of household survey data. Lancet. 2006 Oct 14;368(9544):1357-64. doi: 10.1016/S0140-6736(06)69560-3. PMID 17046468
- [Background] Fernald LC, Gertler PJ, Neufeld LM. Role of cash in conditional cash transfer programmes for child health, growth, and development: an analysis of Mexico's Oportunidades. Lancet. 2008 Mar 8;371(9615):828-37. doi: 10.1016/S0140-6736(08)60382-7. PMID 18328930
- [Background] Grantham-McGregor SM, Powell CA, Walker SP, Himes JH. Nutritional supplementation, psychosocial stimulation, and mental development of stunted children: the Jamaican Study. Lancet. 1991 Jul 6;338(8758):1-5. doi: 10.1016/0140-6736(91)90001-6. PMID 1676083
- [Background] Hamadani JD, Huda SN, Khatun F, Grantham-McGregor SM. Psychosocial stimulation improves the development of undernourished children in rural Bangladesh. J Nutr. 2006 Oct;136(10):2645-52. doi: 10.1093/jn/136.10.2645. PMID 16988140
- [Background] Nahar B, Hossain MI, Hamadani JD, Ahmed T, Huda SN, Grantham-McGregor SM, Persson LA. Effects of a community-based approach of food and psychosocial stimulation on growth and development of severely malnourished children in Bangladesh: a randomised trial. Eur J Clin Nutr. 2012 Jun;66(6):701-9. doi: 10.1038/ejcn.2012.13. Epub 2012 Feb 22. PMID 22353925
- [Background] Tofail F, Hamadani JD, Mehrin F, Ridout DA, Huda SN, Grantham-McGregor SM. Psychosocial stimulation benefits development in nonanemic children but not in anemic, iron-deficient children. J Nutr. 2013 Jun;143(6):885-93. doi: 10.3945/jn.112.160473. Epub 2013 Apr 24. PMID 23616511
- [Background] Gardner JM, Powell CA, Baker-Henningham H, Walker SP, Cole TJ, Grantham-McGregor SM. Zinc supplementation and psychosocial stimulation: effects on the development of undernourished Jamaican children. Am J Clin Nutr. 2005 Aug;82(2):399-405. doi: 10.1093/ajcn.82.2.399. PMID 16087985
- [Background] Fernald LC, Gertler PJ, Neufeld LM. 10-year effect of Oportunidades, Mexico's conditional cash transfer programme, on child growth, cognition, language, and behaviour: a longitudinal follow-up study. Lancet. 2009 Dec 12;374(9706):1997-2005. doi: 10.1016/S0140-6736(09)61676-7. PMID 19892392
- [Background] Robertson L, Mushati P, Eaton JW, Dumba L, Mavise G, Makoni J, Schumacher C, Crea T, Monasch R, Sherr L, Garnett GP, Nyamukapa C, Gregson S. Effects of unconditional and conditional cash transfers on child health and development in Zimbabwe: a cluster-randomised trial. Lancet. 2013 Apr 13;381(9874):1283-92. doi: 10.1016/S0140-6736(12)62168-0. Epub 2013 Feb 27. PMID 23453283
- [Background] Nahar B, Hamadani JD, Ahmed T, Tofail F, Rahman A, Huda SN, Grantham-McGregor SM. Effects of psychosocial stimulation on growth and development of severely malnourished children in a nutrition unit in Bangladesh. Eur J Clin Nutr. 2009 Jun;63(6):725-31. doi: 10.1038/ejcn.2008.44. Epub 2008 Sep 3. PMID 18772893
- [Derived] Hossain SJ, Roy BR, Salveen NE, Hasan MI, Tipu SMMU, Shiraji S, Tofail F, Hamadani JD. Effects of adding psychosocial stimulation for children of lactating mothers using an unconditional cash transfer platform on neurocognitive behavior of children in rural Bangladesh: protocol for a cluster randomized controlled trial. BMC Psychol. 2019 Mar 5;7(1):13. doi: 10.1186/s40359-019-0289-9. PMID 30836984